CLINICAL TRIAL: NCT04824638
Title: A Phase II Trial Assessing Immunogenicity and Safety of COVID-19 mRNA Vaccine BNT162b2 in Adult Volunteers With no History of SARS-CoV-2 Infection Administered With Two Doses of Vaccine (D1-D29) and in Adult Volunteers With Documented History of SARS-CoV-2 Infection (of More Than 5 Months) Administered With Only One Dose of Vaccine
Brief Title: BNT162b2 Vaccination With 2 Doses in COVID-19 Negative Volunteers and With a Single Dose in COVID-19 Positive Volunteers
Acronym: CoviCompareP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS0002S
Record Dates: First submitted 2021-03-07; First posted 2021-04-01 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Immunization; Infection
Keywords: BNT162b2 vaccine; elderly; SARS CoV-2 infected participants
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Participants of group 1 will receive two administrations of BNT162b2 at Day1 and Day29 then at Month8 Participants of group 2 will receive one administration of BNT162b2 at Day1, then at Month8
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: SARS-CoV-2 naive participants (Experimental): participants without antecedent of SARS-CoV-2 infection
  Interventions: Biological: 3 doses of BNT162b2 vaccine
- Group 2: Previously SARS CoV-2 infected participants (Experimental): participants with antecedent of SARS-CoV-2 infection (more than 5 months)
  Interventions: Biological: 2 dose of BNT162b2 vaccine

INTERVENTIONS:
Biological: 3 doses of BNT162b2 vaccine — Administration of BNT162 b2 vaccine (30µg in 0.3mL) at D1 D29 and M8, intramuscularly (participants without antecedent of SARS-CoV-2 infection)
  Arms: Group 1: SARS-CoV-2 naive participants
Biological: 2 dose of BNT162b2 vaccine — Administration of BNT162 b2 vaccine (30µg in 0.3mL) at D1 and M8, intramuscularly (participants with antecedent of SARS-CoV-2 infection)
  Arms: Group 2: Previously SARS CoV-2 infected participants

SUMMARY:
As previously shown, individuals who experienced COVID-19 have developed some protective immunity to reinfection. The magnitude and duration of protection from reinfection conferred by the infection may be weaker after an asymptomatic infection as it is after a symptomatic COVID-19 episode. Moreover, it is known that immunity decreases among older adults compared to younger individuals often referred to as ''immune senescence,'' and leading to a decreased efficacy of vaccination.

This study raises the question of whether a single administration of BNT162b2 in participants with prior SARS-CoV-2 infection leads to sufficient and durable immune response.

We propose to evaluate the level of the single BNT162b2 vaccine dose response according to the severity of the previous SARS-CoV-2 infection in young and elderly participants with the same immunogenicity analyses to assess this response in participants receiving the two-dose vaccination regimen.

DETAILED DESCRIPTION:
This is a national open phase II trial, assessing the immunogenicity and safety of vaccine candidate Pfizer - BNT162b2 against SARS-CoV-2 in participants with no history of SARS-CoV-2 infection receiving two doses of vaccine and in participants with history SARS-CoV-2 infection of more than 5 months and receiving only one dose of vaccine.

A total of 300 volunteers will be included and vaccinated in 2 groups:

Group 1: Adults with no history of SARS-CoV-2 infection(N=150)

* Sub-group 1A: 18 - 45 years old: 50 volunteers
* Sub-group 1B: 65 - 74 years old: 50 volunteers* (minimum of 45)
* Sub-group 1C: At least 75 years old: 50 volunteers* (minimum of 45)

Group 2: Adults with history of SARS-CoV-2 infection of more than 6 months (N=150)

* Sub-group 2A: 18 - 45 years old: 50 volunteers
* Sub-groupe 2B : 65 ans et plus: 100 participants

Within each subgroup of the group 2, a distribution will be respected including:

* 1/3 volunteers with asymptomatic COVID-19 infection,
* 1/3 volunteers with mild COVID-19 infection ((symptomatic but not hospitalized or hospitalized but no oxygen required) and
* 1/3 volunteers with severe COVID-19 infection (hospitalization and oxygen required).

Participants within the group 1 will receive BNT162b2 (Comirnaty®) intramuscularly as a 2-dose series spaced 28 days apart at a dose of 30 µg each, then a booster dose (30µg) at M8.

Participants within the group 2 will receive BNT162b2 intramuscularly as a single dose of 30 µg, then a booster dose (30µg) at M8.

Analyses of humorale and saliva immune responses will be performed in differents centralized laboratories blinded for the trial group, by ELISA at Day -6/D0 (pre-vaccination sample), D29, D57, M6, M12, and M24.

T and B cell analyses will be performed in a sub-group of participants Immunosenescence will be analysed in pre-vaccination samples.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years old or at least 65 years old,
2. Healthy adults or stable medical condition for adults with pre-existing medical conditions. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrolment, nor expected to require any significant change in therapy or hospitalization for worsening disease in foreseeable future.
3. Group 1: Healthy adults with no previous history of SARS COV2 infection (PCR-, antigenic test- or chest TDM- or serology SARS-CoV-2-) Group 2: Healthy adults with history of infection with SARS COV 2 (PCR+, antigenic test+ or chest TDM+ or serology SARS-CoV-2 of more than 5 months) OR have been a household contact subject and have presented COVID-19 symptoms [Experienced at least TWO of the following systemic symptoms: Fever (≥ 38ºC), chills, myalgia, headache, sorethroat, new olfactory and taste disorder(s), gastrointestinal symptoms (diarrhea and/or vomiting) or at least ONE of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, OR clinical or radiographical evidence of pneumonia] since at least 5 months ago and have had a positive SARS-CoV-2 serology between this episode and pre-inclusion.
4. A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

   * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile. OR
   * Is of childbearing potential and agrees to use an effective contraceptive method from at least 4 weeks prior to vaccination until at least 4 weeks after the last vaccination. A participant of childbearing potential must have a negative blood pregnancy test at enrolment visit.
5. Understands and agrees to comply with the study procedures (visits, phone calls) based on Investigator judgement
6. Written and informed consent signed by the person and the investigator (no later than the day of pre-inclusion and prior to any examination realized in the frame of the trial) (article L1122-1-1 of the Public Health Code)
7. Affiliated or beneficiary of a social security scheme (article L1121-11 of the Public Health Code) (AME is not a social security scheme)
8. who agrees to be registered in the national file of persons who lend themselves to biomedical research (article L1121-16 of the Public Health Code).

Exclusion Criteria:

1. Participant is ill or febrile (body temperature ≥ 38.0°C) within 72 prior hours or and/or symptoms suggestive of COVID-19 or being contact subject within the past 14 days at enrolment visit.

   (Ill or febrile participants may be re-scheduled within the trial inclusion period when no longer presenting symptoms, except if condition is COVID19)
2. Participants with positive PCR, antigenic test or chest TDM or serology to SARS-CoV-2 at the enrolment visit, only for the group1.
3. Participants who already received another anti-SARS-CoV-2-vaccine
4. Participants who received BCG given within the last year.
5. Use of immunosuppressive drugs like e.g. corticosteroids at a dosage > 10mg equivalent prednisone /day (excluding topical preparations and inhalers) within 3 months prior to enrolment or 6 months for chemotherapies
6. Received immunoglobulin or other blood product within 3 months prior to enrolment or planned receipt of immunoglobulin or a blood product through study completion.
7. Received any vaccination within 4 weeks prior to first injection or plan to receive a licensed vaccine within 4 weeks after the last injection.
8. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as rash, respiratory difficulty, laryngeal oedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the anti-SARS-CoV-2-vaccine.
9. History of severe allergic event
10. Known HIV, active HCV or HBV infection
11. Any pathological condition, such as cancer, which may be susceptible of reducing immunity response
12. Any bleeding disorder considered as contraindication to intramuscular injection or phlebotomy
13. The use of investigational Ig, investigational monoclonal antibodies or convalescent serum are not allowed during the study
14. Any condition which in the opinion of the investigator may interfere with the aim of the study
15. Pregnant or breastfeeding or positive pregnancy blood test at enrolment visit.
16. An immediate family member or household member of study staff.
17. Participation in another investigational clinical study (Jardé 1 or Jardé 2) within 4 weeks before the enrolment visit or still in an exclusion period from another clinical trial or participation in another investigational clinical study planned before the study completion.
18. People under legal protection measure (tutorship, curatorship or safeguard measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
IgG humoral response to vaccine 28 days post vaccination | at Day 57 for patients of the group1 and at Day 29 for patient of the group 2
  Anti SARS-CoV-2 Spike IgG (ELISA test) 28 days after the last injection i.e. at Day 57 in adult volunteers receiving 2 vaccine doses (group 1, without documented history of SARS-CoV-2 infection) and at Day 29 in adult volunteers receiving 1 vaccine dose (group 2, with documented history of SARS-CoV-2 infection).

SECONDARY OUTCOMES:
humoral response to vaccine | Day 1, Day 29, Day 57, Month 6, Month 8, Month 8+3days, Month 8+15days, Month 8+28 days, Month 8+6 month, Month 24
  Anti SARS-CoV-2 specific IgG at Day1, Day29 (group1), Day57 (group2), [Month8, Month8+3days*, Month8+15 days*, Month8+28 days (participants (*50%)having received the additional vaccine dose)], Month 6, Month8+6months and Month24. Anti SARS-CoV-2 IgA and IgM at Day1, Day29, Day57, Month6, Month8+6months and Month24 (all participants); Month8, Month8+28days (participants that received the additional vaccine dose).Specific neutralizing antibody to SARS-CoV-2 (all participants) and its variants (30 participants per group) by classical in vitro neutralisation assay at Day1, Day29, Day57, Month6, Month8+6months, Month24; Specific neutralizing antibody to SARS-CoV-2 at Month8, Month 8+3days*, Month8+15days* and Month8+28days (participants (*50%) that received the additional vaccine dose). Specific neutralizing antibody to SARS-CoV-2 at day1, Day29, Day57, Month6, Month8+6months, Month24) (all participants). Specific neutralizing antibody to SARS-CoV-2 variants (30 participants per group
T cells response to vaccine | Fluorospot assays : Day 1, Day 29, Day 57, Month 6, Month 8+6months, Month 24 (all participants) and at Month 8, Month 8+28days (participants having received the additional vaccine dose). Phenotyping of antigen specific T-Cells : Day 1 and Month 24
  Fluorospot assays (TH1, TH2, TH17, Cytotoxicity) Phenotyping of antigen specific T-Cells via Mass cytometry at Day 1 and Month24 selected from results of Fluorospot assay
Mucosal response to vaccine | Day 1, Day29, Day57, Month6, Month12, Month24 (all participants) [and Month 8, Month 8+28days, Month 8+6months (participants having received the additional vaccine dose)]
  Mucosal SARS-CoV-2 -specific antibody via measure of IgA, IgM and IgG in saliva by specific home-made and commercially available ELISA assays for salivary IgA and IgG
B cell response to vaccine | Determination of the epitope profiling and B Elispots: Day1, Day57 and Month24. Determination of the B cell repertoire: Day1, Day57 [and Month8, Month8+28days (participants selected for this analysis and having received an additional dose of vaccine]
  Determination of the epitope profiling and B Elispots as well as B cell repertoire (stereotype clonotype) of the humoral response
predictive determinants of vaccine response | at screening visit : (Day -6) and at the latest day (Day 0) before the inclusion visit (Day 1)
  Pre-existing serology for SARS-CoV-2 or other coronavirus, clinical profile of COVID 19 for group 2, immunosenescence profile, transcriptomic analysis, immune cell phenotype
Safety of BNT162b2 vaccine | through 28 days after each dose of vaccine for reactions; throughout the study period (27 months) for others adverse events
  All grade adverse reactions:
  * Immediate reactogenicity defined as any adverse reactions
  * Local and systemic reactogenicity, all grade, measured by solicited adverse reactions
  * Unsolicited adverse reactions
  Others adverse events:
  * Any AEs of grade ≥ 2, .
  * AEs leading to withdrawal .
  * Medically significant AEs
  * SAEs
SARS-CoV-2 infection | during study period (27 months)
  Occurrence of confirmed SARS-CoV-2 infection.
Immunological parameters | at the time of the infection to SARS Cov-2 during study period (27 months)
  Specific neutralizing antibody to SARS-CoV-2 ; Anti SARS-CoV-2(specific to RBD) by Elisa ; Mucosal SARS-CoV-2 -specific antibody via measure of IgA and IgM in saliva ( ELISA test and specific ultrasensitive test); Fluorospot T cell assays.

CONTACTS AND LOCATIONS:
Overall Officials: LEFEBVRE Maeva, MDPhD, Principal Investigator — CIC1413, Hôtel Dieu - CHU Nantes
Locations (11):
- France (11):
  - CIC1412, CHRU Brest, Brest
  - Centre de Recherche Clinique, CHU Côte de Nacre, Caen
  - CIC 1405 , CHU Clermont-Ferrand, Clermont-Ferrand
  - CIC1430, Hôpital Henri Mondor, Créteil
  - CIC1413 , Hôtel Dieu - CHU Nantes, Nantes
  - Service des maladies infectieuses, CHU de Caremeau, Nîmes
  - CIC1417, hôpital Cochin, Paris
  - CIC 1427, Hopital Saint-Louis, Paris
  - URCI, Hôpital Lyon Sud, Pierre-Bénite
  - CIC1434, Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CIC1415, CHRU Tours Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Undecided